CLINICAL TRIAL: NCT02601040
Title: Phase IV Clinical Trial to Assess the Safety, Immunogenicity,Three-year Immune Persistence of Inactivated Hepatitis A Vaccine (HAV) and Live Attenuated HAV Vaccine in Health Chinese Children and Adult
Brief Title: Immunogenicity and Safety of Inactivated and Live Attenuated Hepatitis A Vaccines
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Collaborators: Institute of Medical Biology, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: JSEPI-004
Record Dates: First submitted 2015-10-25; First posted 2015-11-10 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-10

CONDITIONS: Hepatitis A
Keywords: Safety; Immunogenicity; Vaccine; Hepatitis A
MeSH Terms: conditions — Hepatitis A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Attenuated Hepatitis A Vaccine, H2 Strain (Experimental): Health subjects received attenuated Hepatitis A vaccine intramuscularly in the deltoid region.
  Interventions: Biological: Attenuated Hepatitis A Vaccine, H2 Strain
- Inactivated Hepatitis A Vaccine, Lu8 Strain (Experimental): Health subjects received inactivated Hepatitis A vaccine intramuscularly in the deltoid region.
  Interventions: Biological: Inactivated Hepatitis A Vaccine, Lu8 Strain
- Group A Meningococcal Polysaccharide vaccine (Placebo Comparator): Health subjects received Group A Meningococcal Polysaccharide vaccine intramuscularly in the deltoid region.
  Interventions: Biological: Group A Meningococcal Polysaccharide vaccine

INTERVENTIONS:
Biological: Attenuated Hepatitis A Vaccine, H2 Strain — 6.50 lgCCID50/ml in babies aged 18-35 months\6.50 lgCCID50/ml in children aged 3-16 years \6.50 lgCCID50/ml in adults aged 17 up to 65 years old
  Arms: Attenuated Hepatitis A Vaccine, H2 Strain
Biological: Inactivated Hepatitis A Vaccine, Lu8 Strain — 320EU/Vial in babies aged 18-35 months \320EU/Vial in children aged 3-16 years \640EU/Vial in adults aged 17 up to 65 years old\boost at month 6\two-dose
  Arms: Inactivated Hepatitis A Vaccine, Lu8 Strain
Biological: Group A Meningococcal Polysaccharide vaccine — 30µg Group A Meningococcal Polysaccharide vaccine in subjects aged 18 months-65 years old
  Arms: Group A Meningococcal Polysaccharide vaccine

SUMMARY:
The main purpose of this study was to evaluate the safety and immunogenicity of Immunogenicity of Inactivated and Live Attenuated Hepatitis A Vaccines for healthy Chinese people.

ELIGIBILITY:
Inclusion Criteria:

* Only subjects fulfilling all of the following criteria will be eligible for the study:
* People aged from 18 months to 65 years old.
* The subjects or subjects' guardians are able to understand and sign the informed consent
* The subjects or subjects' guardians allow to comply with the requirements of the protocol
* Subjects with temperature <=37.0°C on axillary setting
* The subjects have signed informed consent already

Exclusion Criteria:

* Subjects will not be eligible for the study if any of the following criteria is met:
* Subject who has a medical history of serious disease including Tumor, autoimmune disease, progressive atherosclerosis diseases or complications of diabetes, chronic obstructive pulmonary disease (copd), kidney disease, congestive heart failure etc.
* Have a history of neurological symptoms or signs
* Have medical history or family history relating to allergies, seizures, epilepsy, brain and spirit etc.
* Suffering from serious chronic diseases
* Suffering from known or suspected of diseases including respiratory diseases, acute infection , mothers have HIV infection, cardiovascular disease, severe hypertension, skin diseases, malignant tumor
* Allergic to any ingredient in research, history of allergies to any vaccination (always), especially for people allergic to high protein food like eggs and milk
* Any prior known or suspected damage or abnormal immune function. As for patients who are treated with immune inhibitors or immune enhancer medicine, accept with immunoglobin, blood products and plasma extraction within 3 months
* Any prior diseases including human immunodeficiency virus infection or related
* Bleeding constitution or prolong bleeding time situation
* Accept hepatitis A vaccination within a month
* Received vaccines, other immune globulin, any research drug injections in the past 4 weeks
* People who had any acute illness, needed systemic antibiotics or antiviral treatment in the past 7 days
* Caught a fever with axillary temperature 38°C or higher in past 3 days
* Take part in another clinical researchers
* Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent
* Pregnancy test result is positive

Ages: 18 Months to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 13500 (Actual)
Dates: Start 2011-11; Primary Completion 2014-06 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Changes of hepatitis A antibody concentration | 37 months
  Changes of anti Hepatitis A antibody geometric mean concentrations at pre-vaccination, month 1,12, 24, 36, and 1 months after the booster vaccination.

SECONDARY OUTCOMES:
Incidence of adverse events | 28 days
  Compare incidence of all the solicited events(AEs), unsolicited AEs and serious AEs within 28 days post-vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Jingsi Yang, PhD, Study Chair — Institude of Medical Biology, Chinese Academy of Medical Sciences; Fubao Ma, Study Director — Jiangsu Provincial Center for Disease Control and Prevention; Qiangming Sun, PhD, Principal Investigator — Institude of Medical Biology, Chinese Academy of Medical Sciences; Guodong Kang, Principal Investigator — Jiangsu Provincial Center for Disease Control and Prevention
Locations (2):
- China (2):
  - Jiangsu Provincial Center for Disease Control and Prevention, Nanjing, Jiangsu
  - Institute of Medical Biology -Chinese Academy of Medical Sciences, Kunming, Yunnan

REFERENCES:
- [Derived] Wang X, Luo J, Ma F, Kang G, Ding Z, Pan Y, Zhao Y, Chen J, Feng K, Yan L, Zhang J, Li L, Lan Q, Li D, Yang X, Li G, Yang J, Sun Q. The Safety, Immunogenicity, and Immunopersistence of Hepatitis A Vaccine in HBs-Ag-Positive Participants: A Retrospective Study. Front Cell Infect Microbiol. 2021 Jun 17;11:672221. doi: 10.3389/fcimb.2021.672221. eCollection 2021. PMID 34222044